CLINICAL TRIAL: NCT02951442
Title: Identification of Markers (Klotho-FGF23 Axis) as Determinant in the Evolution of Arterial Stiffness During the First Year of Renal Transplant
Acronym: KLOTHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010/26; 2010-A00413-36 (Other: ANSM)
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2017-01

CONDITIONS: Renal Transplant
Keywords: Arterial stiffness; Klotho-FGF23

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Transplant (Experimental)
  Interventions: Biological: Biological sample; Procedure: Non invasive Arterial investigations; Procedure: Abdominal tomodensitometry

INTERVENTIONS:
Biological: Biological sample
Procedure: Non invasive Arterial investigations
Procedure: Abdominal tomodensitometry

SUMMARY:
The primary objective is to show that the contribution of Klotho by the renal graft is an independent determinant of the evolution of the recipient's central arterial stiffness during the first year of renal transplant. The contribution of Klotho by the graft will be estimated by: its circulating concentrations assay, its urinary excretion assay, and, indirectly, by the circulating concentrations of FGF23. The recipient's central arterial stiffness will be estimated by the measure of the carotid-femoral pulse wave velocity, noninvasive reference method for measuring aortic stiffness in human.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman 18 to 70 years old
* Renal transplant
* Dead donor or alive donor
* Immunosuppression including a calcineurin inhibitor
* Written consent

Exclusion Criteria:

* MultipleTransplant
* Morbid Obesity (Body Mass Index (BMI)> 40 kg/m2 sc)
* Cardiac Arrhythmia
* Lower limbs occlusive arterial disease
* Impossibility to understand the information form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01-28 (Actual); Study Completion 2014-01-28 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral pulse wave velocity | 12 months

SECONDARY OUTCOMES:
Sectional carotid stiffness | 12 months
Carotid intima-media thickness | 12 months
Endothelial function | 12 months
Arterial calcification | 12 months
Pulsed central veinous pressure | 12 months
Klotho concentration | 1 day
FGF23 concentration | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delahousse, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - AH-HP Hôpital Necker enfants malades, Paris
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No